CLINICAL TRIAL: NCT03053934
Title: Evaluation of Online Video Counselling
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Trial no longer feasible
Sponsor: Swinburne University of Technology (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OVC-2016
Record Dates: First submitted 2016-12-21; First posted 2017-02-15 (Actual); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Videoconferencing
Keywords: Online counselling

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional in-person (Active Comparator): Participants randomised to this arm will receive traditional in-person counselling (i.e., treatment will be conducted with the client and clinician occupying the same physical location/room)
  Interventions: Behavioral: Traditional in-person counselling
- Online counselling (Experimental): Participants randomised to this arm will receive treatment from a clinician via videoconferencing (i.e., communication between the client and clinician will occur via webcam)
  Interventions: Behavioral: Online video-based counselling

INTERVENTIONS:
Behavioral: Online video-based counselling — Videoconferencing facilitates communication between individuals (i.e., the counsellor and the client) in different geographical locations enabling them to interact simultaneously with each other on a computer monitor in real time. In other words, both the client and the therapist communicate live using both visual and audio aids simulating in-person therapy albeit from two separate geographical locations.
  Arms: Online counselling
Behavioral: Traditional in-person counselling — Traditional in-person counselling is often referred to as "face-to-face" and can be loosely defined as any mental health intervention, whereby the clinician is in the same room with a client. The terms "in-person" and "same room" are used less frequently, but it has been argued that these terms are more descriptive (since in videoconferencing, clients are also seen "face-to-face" on screen). Therefore, the current study uses the term "in-person" to describe traditional, face-to-face counselling.
  Arms: Traditional in-person

SUMMARY:
The objective of the study is to establish whether online video counselling is at least equally acceptable and equally as effective to clients and clinicians of the Veterans and Veterans Families Counselling Service (VVCS) as in-person counselling. If this is confirmed by the evaluation then online video counselling can be made more widely available to support the veteran and ex-service community, especially for those who may otherwise be unable to attend therapy and for clients who would prefer such web-based services over in-person sessions.

ELIGIBILITY:
Inclusion Criteria:

* Currently residing in Australia
* Eligible to receive support from the Veterans and Veterans Families Counselling Service (VVCS)
* Aged between 18 and 65
* Home access to broadband internet
* Own a device (e.g., computer, laptop, or tablet) that has a webcam and can support videoconferencing
* Be able to reasonably travel to a VVCS centre to access counselling
* Referred for one-to-one counselling or therapy
* Be willing and able to receive either modality of treatment (i.e., online or in-person counselling).

Exclusion Criteria:

* Not currently residing in Australia
* Not eligible to receive support from VVCS
* Significant current risk issues or levels of acute distress requiring crisis management
* Current serving member of the Australian Defence Force with a high security clearance (above Baseline Vetting)
* Referred for couple or family counselling.
* Have received a psychiatric diagnosis of post-traumatic stress disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Group x Time Interaction for overall mental health as measured by the K10 from baseline to 16-week follow up | Baseline, 8-week follow-up, 16-week follow-up
  0 to 16 week difference in K10 scores in group x time interaction. The Kessler Psychological Distress Scale (K10) (Kessler et al., 2002) is a 10-item questionnaire intended to yield a global measure of distress based on questions about anxiety and depressive symptoms that a person has experienced in the most recent 4-week period.

SECONDARY OUTCOMES:
Group x Time Interaction for the Outcome Rating Scale from baseline to 16-week follow up | Baseline, 8-week follow-up, 16-week follow-up
  0 to 16 week difference in ORS scores in group x time interaction. The Outcome Rating Scale (ORS, Miller, Duncan, Brown, Sparks, & Claud, 2003) will also be administered at all three time points. This is a 4-item self-report inventory that measures three different dimensions of client functioning generally considered as valid indicators of treatment progress: individual (or symptomatic) functioning, interpersonal relationships, and social role performance (work adjustment, quality of life).
Group x Time Interaction for Quality of Life from baseline to 16-week follow up | Baseline, 8-week follow-up, 16-week follow-up (only administered to participants completing the survey online)
  0 to 16 week difference in AQoL-8D scores in group x time interaction. The Assessment of Quality of Life-8D (AQoL-8D, Richardson et al., 2014) is a 35-item measure of health related quality of life which is sensitive to mental health issues, and is suitable for calculation of QALYs.
  This measure is to be administered at all three data collection points, however, due to the length of this measure, it would be too time consuming for participants to complete this measure over the telephone. Therefore, this measure will only be completed by participants who complete the assessment online.
Therapeutic (or Working) Alliance | 8-week follow up
  The Working Alliance Inventory - Short Revised (WAI-SR). This is a 12-item form of the WAI (Horvath & Greenberg, 1989). It is a self-report inventory that measures the quality of the therapeutic relationship from the client's perspective.
Client Satisfaction | 8-week follow up
  The NHS Friends and Family Test (FFT). This is a single-item measure used to help service providers understand whether their clients are satisfied with the service provided.
Client and Clinician Experiences | Up to 6 months post-treatment
  Semi-structured interviews will also be conducted on clients and clinicians to further investigate their respective experiences with the form of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Denny Meyer, Principal Investigator — Swinburne University of Technology
Locations (1):
- Swinburne University of Technology, Hawthorn, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Undecided